CLINICAL TRIAL: NCT02270294
Title: Acute Effects of Thai Traditional Massage on Cerebrovascular Reactivity in Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr.Daroonwan Suksom, DSuksom, Chulalongkorn University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SPSC-3
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Thai traditional massage; Vascular function; Cerebral blood flow; Cerebrovascular reactivity
MeSH Terms: conditions — Ischemic Stroke | interventions — Medicine, Thai Traditional

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Thai traditional massage (Experimental)
  Interventions: Other: Thai traditional massage
- No massage (Sham Comparator)
  Interventions: Other: No massage

INTERVENTIONS:
Other: Thai traditional massage — Thai traditional massage treatment based on original Thai traditional massage at Wat Po was use in this study. The participants will be assigned to receive one time of Thai traditional massage one time. Thai traditional massage techniques consists of petrissage, friction, and passive stretching on head, neck, shoulders, arms, back and legs for 60 minutes.
  Other Names: Thai massage
  Arms: Thai traditional massage
Other: No massage — The participants will be asked to lie down in relaxant position on bed without sleep for 60 minutes.
  Arms: No massage

SUMMARY:
The investigators hypothesize that Acute Thai traditional massage will yield beneficial effects on cerebrovascular reactivity in ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. A single ischemic stroke with Middle cerebral artery (MCA) stenosis
2. Men or women age 50-80 years
3. Physician's approvals to participate the study
4. Stroke experienced at least 7 days of ischemic stroke onset and no more than 6 months before study enrollment
5. The modified rankin scale level is 2 or 3

Exclusion Criteria:

1. History of serious diseases

   * Musculoskeletal diseases (Chronic arthritis, Lower spondylosis/spondylolisthesis with radiculopathy, Spinal deformity, Cervical spondylosis, Rheumatoid arthritis)
   * Cardiovascular diseases (Poorly control hypertension, Heart disease class C and D)
   * Neurological disorders (Peripheral neuropathy, Parkinson)
   * Respiratory diseases (Chronic Obstructive Pulmonary Disease)
   * Brain disorders (Cardioembolic, Severe dementia, Alzheimer's disease)
   * Medical condition precluding taking Anticoagulant and Statin drug
2. Temporal window were not found

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2016-08-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cerebrovascular reactivity | baseline, Post-test (immediately: 0 min after finish massage intervention, 60 min, 120 min, 24 Hrs.
  - Cerebrovascular reactivity or cerebral CO2 reactivity test will be assessed using the ultrasound equipment (CX50, Philips, USA). Blood flow velocity (BFV) of the middle cerebral artery (MCA) will be measured during normocapnic, hypocapnic, and hypercapnic states. Subjects will be asked to wear nose clips and breathe only through a mouthpiece. Baseline (3 minutes) recordings will be taken during spontaneous breathing of room air and then subjects underwent 1 minute of maximal voluntary hyperventilation with a duty cycle of 1 second. The MCA-BFV will be recorded during the last 20 seconds of hyperventilation. After that, subjects will be asked to breathe air containing a mixture of 5 % CO2 and 21 % O2 balanced with nitrogen spontaneously for 3 minutes and the MCA-BFV will be recorded during the last minute of hypercapnia.

SECONDARY OUTCOMES:
Change from baseline in stress indicators | Baseline, Post-test (immediately: 0 min after finish massage intervention)
  - Serum cortisol will be measured with cortisol EIA kit (Enzo Life Science, Switzerland).
Change from baseline in stress indicators | Baseline, Post-test (immediately: 0 min after finish massage intervention, 60 min, 120 min, 24 Hrs.
  - Heart rate variability (HRV) will be measured using the Heart rate monitoring (RS800CX, Polar Electro, Oy, Finland)
Change from baseline in Peripheral arterial stiffness | Baseline, Post-test (immediately: 0 min after finish massage intervention, 60 min, 120 min, 24 Hrs.
  - Pulse wave velocity measurement will be assessed with MD6 bidirectional transcutaneous Doppler probe (Hokanson, Bellevue, WA, USA). All subjects will be monitored with an EKG and PWV measurements in the computer and used as timing markers for PWV identification.
Change from baseline in blood chemistry | baseline, Post-test (immediately: 0 min after finish massage intervention)
  * Nitric oxide (NO) will be measured in plasma samples with Colorimetric nitric oxide assay kit (Biovision, USA).
  * Beta-endorphin will be measured in serum samples with the commercial assay kit (Beta-endorphin [bEP] BioAssay ELISA kit [Human], US Biological Life Science).
  * Malondialdehyde (MDA) will be determined using thiobarbituric acid reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathumwan, Bangkok, Thailand